CLINICAL TRIAL: NCT04194229
Title: Use of Cytoflavin Solution at the Time of Early Rehabilitation in Patients With Post-intensive Care Syndrome Who Underwent Ischemic Stroke
Brief Title: Cytoflavin in the Rehabilitation of Post-intensive Care Syndrome in Stroke Survivors
Status: Completed | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-C
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke; Post Intensive Care Unit Syndrome
Keywords: Ischemic stroke; Post-intensive care syndrome; Cytoflavin; Rehabilitation; Metabolograph; Utilization O2; Verticalization
MeSH Terms: conditions — Ischemic Stroke; postintensive care syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group 1: Patients that receive Cytoflavin® medication i/v drop infusion at a dose of 10 ml of solution for injection per 200 ml of 0.9 % sodium chloride solution for 10 days in addition to a set of neurorehabilitation activities
- Group 2: Patients that subjected to the standard set of neurorehabilitation activities for 10 days without being prescribed Cytoflavin® medication

SUMMARY:
Objective - to assess the effect of Cytoflavin® and its tolerability within the integrated program of rehabilitation of patients who underwent ischemic stroke

DETAILED DESCRIPTION:
Cerebral stroke (CS) remains one of the key issues of modern society, being a predominant cause of deep and persistent disability of the population. Huge social and economic damage arising from cerebrovascular diseases raises the problem of improving medical care for strokes among the most relevant scientific and practical tasks of neurology Regulation of energy metabolism is considered a powerful tool for acute conditions relief, including those that occur due to acute impairment of cerebral blood flow. A number of adjuvant energy protector concomitant medications with systemic pharmacodynamic properties based on signaling (hormonal) and substrate mode of action of succinic acid and other mitochondrial substrates and co-factors was created for this A significant role in the rehabilitation of patients who underwent CS is assigned to the treatment of complications of care in the intensive care unit, the so-called post-intensive care syndrome (PICS), which is a set of somatic, neurological, social and psychological consequences of periods in intensive care unit (ICU) conditions that bring limitations to the patient's daily activities In the Brain Institute Clinic (Ekaterinburg), the first results of the metabolic status monitoring during physical and cognitive exercise in patients with PICS were obtained. These results prove that control over metabolic state holds the promise of developing approaches to increasing exercise tolerance Taking into account the effectiveness of Cytoflavin® in treatment of acute impairment of cerebral circulation and consequences of cerebrovascular diseases, on the one hand, and its classification as a metabotropic energy corrector, on the other hand, the evaluation of Cytoflavin® medication tolerability in the integrated program of neurorehabilitation of patients with PICS after ischemic stroke presents a significant interest.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and above;
* Patients who underwent ischemic stroke;
* The period from the development of ischemic stroke is not less than 12 and not more than 28 days;
* Staying in intensive care unit for no less than 72 hours;
* Diagnosed post-intensive care syndrome (PICS);
* Functional status assessed using the modified Rankin scale amounts to 4-5;
* Gravity gradient of 20° to 40° upon inclusion in observational non-interventional program

Exclusion Criteria:

* Vegetative state;
* Mechanical ventilation lasting more than 72 hours after the development of ischemic stroke;
* Surgical treatment for cerebral stroke (decompressive craniectomy; thromboextraction etc.);
* Premorbid (before the development of ischemic stroke) level of functional activity assessed using the modified Rankin scale amounts to 4 or 5;
* Signs of increasing neurological deficit or enlargement of hypoperfusion zones on CT scans within 24 hours before inclusion in observational non-interventional program;
* Level of consciousness ≤ 5 according to Glasgow Coma Scale and/or ≥ 1 according to Richmond Agitation-Sedation Scale (RASS);
* Behavioral Pain Scale (BPS) or Visual Analogue Scale assessment score of more than > 0 at the moment of inclusion;
* Systolic blood pressure < 90 and > 180 mm Hg;
* Diastolic blood pressure ≥ 110 mm Hg;
* Mean ABP < 60 mm Hg;
* Clinical and/or electrocardiographic signs of acute coronary syndrome (including de novo ST elevation or depression, negative T-waves amplitude formation and buildup, formation of pathological Q-wave, increase in the level of markers of myocardial injury - troponin T or I, creatine phosphokinase-MB, LDH-1), or diagnosed acute myocardial infarction occurring within a month before inclusion in observational program;
* Acute heart arrhythmias;
* Heart rate (HR) < 60 or > 100 per minute;
* Spontaneous respiration rate (RR) < 10 or > 30 per minute;
* Arterial oxygen saturation (SpO2) < 90 %;
* Venous serum glucose level ≤ 4 mmol/L;
* Axillary body temperature ≥ 38.5 °C;
* Hematocrit ≤ 30 %;
* Level of hemoglobin ≤ 80 g/l;
* Serum total protein ≤ 55 g/l;
* Positive passive leg raising test (PRL-test);
* Acute heart failure;
* Acute respiratory failure;
* Acute kidney injury;
* Acute liver cell failure;
* Congestive heart failure;
* Chronic respiratory failure, stage greater than I;
* Chronic kidney disease with estimated glomerular filtration rate using Cockcroft-Gault formula < 60 ml/min/1.73 m2;
* Clinically significant deviations in the results of complete blood count, blood chemistry, common urine analysis, except those that are acceptable according to other non inclusion criteria;
* Purulent-inflammatory diseases at any location;
* Refuse of the patient to undergo verticalization or exercise sessions;
* Use of medicinal products belonging to the pharmaceutical therapeutic category of metabolic drugs at the time of inclusion in observational non-interventional program, as well as plans for their use during study;
* Plans for use of physical rehabilitation methods other than verticalization and cycling exercise sessions during the course of the program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants of the observational program will be male and female adults who underwent ischemic stroke NLT 12 and NMT 28 days before being admitted to the observational program with diagnosed PICS.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Median time to achieving gravity gradient of 90° | 10 days
  Median time (in days) to achieving gravity gradient of 90°.

SECONDARY OUTCOMES:
Proportion of patients who achieved gravity gradient of 90° | 5 and 10 days
  Proportion of patients who achieved gravity gradient of 90° by day 5 and 10 days of rehabilitation activities
Change in of oxygen consumption during 90° verticalization | 5 and 10 days
  Change in of oxygen consumption during 90° verticalization
Change in the Medical Research Council (MRC) scale for muscle strength score | 5 and 10 days
  Medical Research Council scale for muscle power (MRC), where 0 - tetraplegia, 60 - normal value
Change in Barthel index (BI) | 5 and 10 days of rehabilitation activities
  Barthel index (BI), when 0 - complete inability to self-service, 100 - full capability of self-service
Change in Modified Rankin scale (MRS) score | 5 and 10 days of rehabilitation activities
  Modified Rankin scale (MRS), when 0 - no disability, 5 - severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Belkin, Prof, Principal Investigator — Brain Institute Clinic, Yekaterinburg
Locations (1):
- Brain Institute Clinic, Yekaterinburg, Sverdlovsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Belkin AA, Leiderman IN, Kovalenko AL, Rizakhanova OA, Parfenov SA, Sapozhnikov KV. Cytoflavin as a modulator of rehabilitation treatment of patients with ischemic stroke complicated by post-intensive care syndrome. S.S. Korsakov Journal of Neurology and — https://www.mediasphera.ru/issues/zhurnal-nevrologii-i-psikhiatrii-im-s-s-korsakova/2020/10/1199772982020101027
- See also: Belkin AA, Leiderman IN, Kovalenko AL, Rizakhanova OA, Parfenov SA, Sapozhnikov KV. Tsitoflavin kak komponent reabilitatsionnogo lecheniya patsientov s ishemicheskim insul'tom, oslozhnennym PIT-sindromom — https://pubmed.ncbi.nlm.nih.gov/33244954/